CLINICAL TRIAL: NCT06246838
Title: 68Ga PET/CT Versus 99mTc SPECT/CT for Lung Perfusion and Ventilation Scintigraphy; a Technical and Practical Feasibility Study
Acronym: GaTcha
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Arthur Braat, Dr. A.J.A.T. Braat, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GaTcha
Record Dates: First submitted 2024-01-12; First posted 2024-02-07 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Pulmonary Embolism; Ventilation Perfusion Mismatch
Keywords: Ga-68-MAA; Galligas; Tc-99m-MAA; Technegas; PET/CT; SPECT/CT
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ga-68 V/Q PET/CT — Head-to-head comparison of Ga-68 V/Q PET/CT vs Tc-99m V/Q SPECT/CT
  Other Names: Tc-99m V/Q SPECT/CT

SUMMARY:
Lung perfusion scintigraphy with 99mTc-MAA and ventilation scintigraphy with Technegas (V/Q SPECT/CT) has been the cornerstone for the detection of pulmonary embolisms (PE) for many decades. In last two decades after the introduction of pulmonary CTA, general PE detection has shifted towards CTA and V/Q SPECT/CT has become the modality of choice for specific patient populations (iodine contrast allergy, poor kidney function, pregnancy, etc.) or indications (pre-operative risk stratification, chronic embolism detection, pulmonary hypertension). V/Q SPECT/CT acquisition is performed on a gamma camera, but this technique has distinct challenges and/or disadvantages. A potential alternative is the nowadays broadly available. 68Ga as a positron emitter allows PET/CT imaging. Replacing 99mTc with 68Ga in both MAA and aerosol suspension is easy and requires no modifications. However, 68Ga-V/Q with PET/CT will resolve many of the disadvantages of V/Q SPECT/CT. International studies have proven safety and feasibility of replacing 99mTc with 68Ga and preliminary work by international colleagues and our institute have shown validated preparations of the radiopharmaceuticals. However, in our institution, clinical translation is hampered by lack of data on technical acquisition parameters for our scanners. The aim of this small study is to get more insights into technical parameters for image acquisition, logistical feasibility of V/Q PET/CT, and confirm preliminary non-inferiority of this new technique over the current clinical standard (V/Q SPECT/CT).

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥18 years and declared competent
* Provided written informed consent
* Referred to the Nuclear Medicine Department for a conventional V/Q-SPECT/CT
* Indication for conventional V/Q-SPECT/CT includes known or suspected pulmonary embolism

Exclusion Criteria:

- Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Qualitative assessment of V/Q-PET/CT | Study participation is maximum 1 week.
  Qualitative assessment of different image acquisition parameters for V/Q PET/CT, as determined by blinded assessment by experienced nuclear medicine physicians in a 5-point Likert scale of V/Q PET (compared to the clinical reference standard V/Q SPECT).
Quantitative assessment of V/Q PET/CT | Study participation is maximum 1 week.
  Quantitative assessment of different image acquisition parameters for V/Q PET/CT, by comparison semi-quantitative measurements of V/Q PET (e.g. signal-noise ratio's, etc.).

CONTACTS AND LOCATIONS:
Locations (1):
- UMC Utrecht, Utrecht, Netherlands